CLINICAL TRIAL: NCT00781950
Title: A Double Blind, Randomized, Placebo Controlled, Study for Assessment of Dietary Flaxseed on Improving Symptoms of Cardiovascular Disease in Patients With Peripheral Arterial Disease
Brief Title: Effects of Dietary Flaxseed on Symptoms of Cardiovascular Disease in Patients With Peripheral Arterial Disease
Acronym: FLAXPAD
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Dr. Grant Pierce (Other)
Responsible Party: Sponsor-Investigator, Dr. Grant Pierce, Executive Director, Research Enterprise, St. Boniface Hospital
Organization: St. Boniface Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 10941-011
Record Dates: First submitted 2008-10-28; First posted 2008-10-29 (Estimated); Results first posted 2014-12-12 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2016-10

CONDITIONS: Peripheral Arterial Disease
Keywords: PAD; Peripheral Arterial Disease; Diabetes; Atherosclerosis; Flax; Flaxseeds; Functional Foods; Essential Fatty Acids; Winnipeg
MeSH Terms: conditions — Peripheral Arterial Disease; Diabetes Mellitus; Atherosclerosis | interventions — Linseed Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Randomized, Blinded Controlled Arm of patients receiving placebo food products (ie: bagels, muffins, bars, pasta, buns, and milled seeds) containing a mixture of wheat and wheat bran to replace the flaxseed daily for one year.
  Interventions: Dietary Supplement: Placebo
- Flaxseed (Experimental): Randomized, Blinded group of patients that will be given food products (ie: bagels, muffins, bars, pasta, buns, and milled seeds) containing 30 g of milled flaxseed daily for one year
  Interventions: Dietary Supplement: Flaxseed

INTERVENTIONS:
Dietary Supplement: Flaxseed — 30 grams of milled flaxseed per day in food products or on its own.
  Arms: Flaxseed
Dietary Supplement: Placebo — Wheat and Mixed Dietary Oils
  Arms: Placebo

SUMMARY:
This Clinical Trial is being conducted to study how patients with peripheral arterial disease (a condition in which the blood vessels of the extremities are affected) respond to a dietary regimen of flaxseed. The purpose of the study is to examine whether or not dietary flaxseed have any effect on improving symptoms of cardiovascular disease. Additionally, the effects of dietary flaxseed on exercise tolerance will be assessed.

DETAILED DESCRIPTION:
The proposed trial is a one year, double blinded, placebo controlled study designed to examine and compare the effects of dietary ground flaxseed supplementation in volunteers with claudication secondary to lower extremity atherosclerotic arterial disease (peripheral arterial disease). The original proposal was for a two year study duration but this was truncated at one year to insure patient compliance remained high. This patient population is likely to benefit from flaxseed because there is a high prevalence of accelerated atherosclerosis and a higher than normal incidence of arrhythmias, myocardial infarctions and stroke. This study will be focus on whether dietary flaxseed can reduce clinical manifestations of peripheral arterial disease and increase exercise capacity in these patients. Two general hypotheses will be tested in this proposal. First, we hypothesize that fewer primary and secondary events (all-cause mortality, cardiovascular mortality, stroke, myocardial infarctions, angina, arrhythmias) will occur in patients who ingest flaxseed in their diet. Secondly, we hypothesize that dietary flaxseed supplementation will be associated with beneficial effects on exercise performance, blood pressure and circulating lipid levels. This trial will generate data on the safety, tolerability, cardiovascular efficacy and genomic response to a diet rich in flaxseed in patients with peripheral arterial disease (PAD).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with peripheral arterial disease for more than 6 months.
* Male or female with claudication secondary to lower extremity atherosclerotic arterial disease. (with limited IC but not incapacitated for walking on the level) confirmed with ankle/brachial pressures< or = to 0.9 in one or both legs) or who have had a previous intervention for peripheral arterial disease.
* Over 40 years old
* Able to comply with protocol requirements
* Able to provide informed consent
* Subjects taking anti-platelet therapy medication must be on a stable dose for 3 months prior to as well as during the study.
* Subjects taking lipid lowering medication must be on a stable dose for 3 months prior to as well as during the study.

Exclusion Criteria:

* Patients with ischemic rest pain in limbs, ulceration, or gangrene.
* At baseline, any condition that prevents walking on a treadmill.
* History of major bleeding.
* Patients with bowel disease (including Crohn's disease, celiac disease, peptic ulcer disease, irritable bowel syndrome and diverticulosis).
* Patients with an estimated life expectancy less than 2 years and with high baseline cardiac risk (post ischemic or diabetic cardiomyopathy with EF<40%, Canadian Cardiovascular Society Class 3 or 4 angina or need for coronary revascularization procedures).
* Moderate to severe renal failure.
* Subjects that are on supplements other that those prescribed by their clinician for the entire duration of the study.
* Fish limitations (no more than 2 fish meals per week)
* Gluten allergy
* Subjects with allergies to any ingredient in the study product or placebo.
* Patients who plan to undergo surgery during the course of the trial.

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2008-10; Primary Completion 2011-03 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grant Pierce, PhD, Principal Investigator — University of Manitoba

REFERENCES:
- [Derived] Caligiuri SP, Rodriguez-Leyva D, Aukema HM, Ravandi A, Weighell W, Guzman R, Pierce GN. Dietary Flaxseed Reduces Central Aortic Blood Pressure Without Cardiac Involvement but Through Changes in Plasma Oxylipins. Hypertension. 2016 Oct;68(4):1031-8. doi: 10.1161/HYPERTENSIONAHA.116.07834. Epub 2016 Aug 15. PMID 27528063
- [Derived] Edel AL, Rodriguez-Leyva D, Maddaford TG, Caligiuri SP, Austria JA, Weighell W, Guzman R, Aliani M, Pierce GN. Dietary flaxseed independently lowers circulating cholesterol and lowers it beyond the effects of cholesterol-lowering medications alone in patients with peripheral artery disease. J Nutr. 2015 Apr;145(4):749-57. doi: 10.3945/jn.114.204594. Epub 2015 Feb 18. PMID 25694068
- [Derived] Caligiuri SP, Aukema HM, Ravandi A, Guzman R, Dibrov E, Pierce GN. Flaxseed consumption reduces blood pressure in patients with hypertension by altering circulating oxylipins via an alpha-linolenic acid-induced inhibition of soluble epoxide hydrolase. Hypertension. 2014 Jul;64(1):53-9. doi: 10.1161/HYPERTENSIONAHA.114.03179. Epub 2014 Apr 28. PMID 24777981
- See also: Canadian Centre for Agri-food Research in Health and Medicine — http://www.sbrc.ca/ccarm

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Randomized, Blinded Controlled Arm of patients receiving placebo food products (ie: bagels, muffins, bars, pasta, buns, and milled seeds) containing a mixture of wheat, wheat bran, and mixed dietary oils to replace the flaxseed daily for one year.
Period: Overall Study
Arm/Group | Placebo | Flaxseed
Started | 52 | 58
Completed | 41 | 45
Not Completed | 11 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Flaxseed | Total
Number analyzed (Participants) | 52 | 58 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (9.4) | 67.4 (8.06) | 67.3 (8.5)
Gender [Count of Participants; unit: Participants]
  Female | 14 | 15 | 29
  Male | 38 | 43 | 81
Region of Enrollment [Number; unit: participants]
  Canada | 52 | 58 | 110

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With All-cause Mortality, Cardiovascular Mortality, Stroke, and Myocardial Infarctions
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Placebo | Flaxseed
Number analyzed (Participants) | 52 | 58
participants | 4 | 5

2. Secondary Outcome: Effects on Exercise Performance, Blood Pressure and Circulating Lipid Levels.
Time Frame: 1 year
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | Flaxseed
Number analyzed (Participants) | 41 | 45
mmHg
  Final Systolic Blood Pressure | 145.6 (3.4) | 136.2 (3.8)
  Final Diastolic Blood Pressure | 78.5 (1.5) | 71.8 (1.7)

ADVERSE EVENTS:
Description: The adverse events were recorded by the research nurse upon follow-up visits.
Arm/Group | Placebo | Flaxseed
Serious Adverse Events (participants affected / at risk) | 9/52 | 15/58
Other Adverse Events (participants affected / at risk) | 0/52 | 3/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=52) | Flaxseed (N=58)
Increased Claudication (Blood and lymphatic system disorders) | 3 | 7
Iliac Artery Stenosis (Blood and lymphatic system disorders) | 1 | 0
Rest Pain in Limbs (Blood and lymphatic system disorders) | 0 | 2
Increased Numbess in Extremities (Nervous system disorders) | 1 | 0
Ulcerative Cellulitis (General disorders) | 0 | 1
Death (General disorders) | 0 | 1
Stroke (General disorders) | 1 | 3
Myocardial Infarction (Cardiac disorders) | 3 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=52) | Flaxseed (N=58)
Nausea (General disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes